CLINICAL TRIAL: NCT01397331
Title: Influence of Anesthesia on Mechanical Efficiency of Left Ventricle in Patients Undergoing Open Heart Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Technical problems with data acquisition and interpretation; problems with recruitment
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sergey Preisman, M.D., Department of Anesthesia and Intensive Care, Sheba Medical Center, Tel Hashomer, Israel 52621
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-09-7199-SP-CTIL
Record Dates: First submitted 2011-07-14; First posted 2011-07-19 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2011-07

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery; Disorder; Heart, Functional, Postoperative, Cardiac Surgery
Keywords: inhalational anesthesia; intravenous anesthesia; cardiac surgery
MeSH Terms: interventions — Isoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhalational anesthesia (Active Comparator): Group of patients undergoing the surgery under anesthesia based on inhalational anesthetic
  Interventions: Drug: Isoflurane
- TIVA (Active Comparator): Group of patients undergoing the surgery under total intravenous anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Isoflurane — Anesthesia based on inhalation of 1-1.5 Minimal Alveolar Concentration of Isoflurane with the addition of infusion of remifentanil
  Arms: Inhalational anesthesia
Drug: Propofol — Anesthesia based on the infusion of 2-5 mg/kg/h of propofol with the addition of infusion of remifentanil
  Arms: TIVA

SUMMARY:
The aim of the study is to delineate and compare the changes in coupled mechanical properties of left ventricle and arterial vascular bed caused by two popular anesthetic protocols commonly used in cardiac surgery (intravenous, based on the infusion of propofol, versus inhalational, based on isoflurane) on different stages of the surgery.

DETAILED DESCRIPTION:
Background

From mechanical point of view the goal of the cardiovascular system is to distribute the kinetic energy of blood ejection from the left ventricle (LV) to body organs with minimal loss and greatest efficiency. The left ventricle and the arterial circulation work as "coupled" system. The ideal coupling supposes that a maximum of the energy produced by the LV is converted into forward flow to perfuse the body organs. This matching between "the source" (LV) and "the load" (arterial circulation) is governed by the mechanical properties of these parts of cardiovascular system.

Variety of pathological conditions change this coupling in such a way that may adversely affect the organ blood flow in the presence of unchanged or even high cardiac output, or significantly increase the metabolic demand on the LV for the maintenance of adequate systemic perfusion due to decrease of mechanical efficiency of the work produced by LV.

Although effects of anesthetic agents on myocardial contractility and peripheral vascular tone were extensively studied in clinical conditions, little is known about their influence on ventriculo-arterial coupling. Propofol and inhalational agents appear to impair this equilibrium in animal experiments. This is not surprising, since these agents cause complex dose-dependent changes in many physiologic parameters, including myocardial contractility, left ventricular preload and afterload, diastolic properties of myocardium and baroreceptor control of hemodynamics. Although these properties of anesthetic agents have been delineated extensively, very limited data characterizing their influence on ventriculo-arterial coupling in clinical conditions exist. This information is especially meaningful while planning the anesthetic management of patients undergoing cardiac surgery, where maintenance of circulatory homeostasis is of outmost importance. Since the main hemodynamic goal during anesthesia of the patient with cardiovascular disease is to provide optimal tissue perfusion with minimal myocardial oxygen demand, i.e. with maximal mechanical efficiency, knowledge of anesthetic induced changes in ventriculo-arterial coupling is extremely relevant from the clinical point of view.

The most convenient method for the evaluation of ventriculo-arterial coupling is the analysis of the relationship between LV end-systolic elastance, load-independent measure of myocardial contractility, and effective arterial end-systolic elastance, measure mechanical loading conditions8. Physiological data necessary for the calculation of these parameters may be acquired in relatively non-invasive way by combining and analyzing together recording of arterial blood pressure waveform and data of changes of LV volume, which may be obtained by means of echocardiography.

Objectives

General

The aim of the study is to delineate and compare the changes in ventriculo-arterial coupling caused by two popular anesthetic protocols commonly used in cardiac surgery (intravenous, based on the infusion of propofol, versus inhalational, based on isoflurane) on different stages of the surgery.

Specific

1. To compare influence of two anesthetic protocols on myocardial contractility at the end of the surgery.
2. To assess net changes in effective arterial elastance produced by surgery with the use of cardiopulmonary bypass and evaluate possible differences between these two anesthetic protocols in respect to changes of arterial tone.
3. To evaluate the preservation of ventriculo-arterial coupling by two different anesthetic modes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cardiac surgery

Exclusion Criteria:

* Emergent surgery.
* History of previous cardiac surgery.
* Significant arrhythmias.
* More than trivial valvular disorder.
* Absence of written informed consent.
* Contraindications for transesophageal echocardiography.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2012-06-27 (Actual); Study Completion 2012-06-27 (Actual)

PRIMARY OUTCOMES:
Changes of the relationship between left ventricular end-systolic elastance and effective arterial end-systolic elastance. | 15 minutes and 30 minutes after the induction of anesthesia in Inhalational Group and TIVA Group respectively, 15 minutes after the separation from cardiopulmonary bypass, and before the transfer of the patient to the Intensive Care Unit in both groups

SECONDARY OUTCOMES:
Changes in vascular tone and cardiac afterload | 15 minutes and 30 minutes after the induction of anesthesia in Inhalational Group and TIVA Group respectively, 15 minutes after the separation from cardiopulmonary bypass, and before the transfer of the patient to the Intensive Care Unit in both groups
  arterial end-systolic elastance, left ventricular end-systolic stress
Changes of measures of global systolic left ventricular function | 15 minutes and 30 minutes after the induction of anesthesia in Inhalational Group and TIVA Group respectively, 15 minutes after the separation from cardiopulmonary bypass, and before the transfer of the patient to the Intensive Care Unit in both groups
  left ventricular end-systolic elastance, systolic strain and strain rate, myocardial performance index, ejection fraction

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Preisman, M.D., Principal Investigator — Department of Anesthesia and Intensive Care, Sheba Medical Center, Israel 52621
Locations (1):
- Department of Anesthesia and Intensive Care, Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel